CLINICAL TRIAL: NCT06211751
Title: A Phase Ib Clinical Trial to Evaluate the Safety, Efficacy and Pharmacokinetics of TQB3909 Tablets Combined With TQB3702 Tablets in Hematologic Malignancy Subjects.
Brief Title: A Clinical Trial of TQB3909 Tablets Combined With TQB3702 Tablets in Patients With Hematologic Malignancy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-TQB3702-Ib -01
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3909 tablets+ TQB3702 tablets (Experimental): TQB3909 tablets combined with TQB3702 tablets, administered orally, 28 days as a treatment cycle.
  Interventions: Drug: TQB3909 tablets; Drug: TQB3702 tablets

INTERVENTIONS:
Drug: TQB3909 tablets — TQB3909 is a protein inhibitor.
Drug: TQB3702 tablets — TQB3702 is a kinase inhibitor.

SUMMARY:
This is an open, multi-cohort clinical study. The first phase is a dose escalation study and the second phase is a dose expansion study based on the Maximum tolerated dose (MTD) / Recommended Phase II Dose (RP2D) obtained in the first phase. The purpose is to evaluate the safety and preliminary efficacy of TQB3909 tablets combined with TQB3702 tablets in hematologic malignancy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined the study, signed informed consent form, and with good compliance.
* ≥ 18 years old, ≤75 years old (when signing informed consent form); Eastern Cooperative Oncology Group (ECOG) physical status: 0-2; at least 3 months expected survival period.
* Subject population:

  1. Dose escalation stage: non-Hodgkin's B-cell lymphoma;
  2. Dose expansion stage: non-Hodgkin's lymphoma, etc.
* At least 1 lesion / measurable disease for efficacy evaluation.
* The function of main organs is normal.
* Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after the completion of the study; a negative serum pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects; male patients should agree to use contraception during the study period and for at least 6 months after the completion of the study.

Exclusion Criteria:

* Patients has occured or is currently having other malignant tumors within 5 years. The following two conditions can be included: other malignant tumors treated with a single operation to achieved 5 consecutive years of disease free survival (DFS). Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basal membrane)] and papillary thyroid carcinoma.
* Burkitt lymphoma, lymphoblastic lymphoma/leukemia, etc.
* For cohort A and cohort B: Richter transformation occured.
* Subjects with central nervous system (CNS) aggression;
* Previously received allogeneic hematopoietic stem cell transplantation;
* For Cohort B/D/E: Received autologous hematopoietic stem cell transplantation within 3 months before the first dose;
* Multiple factors that affect the absorption of oral medications (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction);
* Unrelieved toxicity of ≥CTCAE grade 1 due to any previous treatment, excluding alopecia and fatigue;
* Major surgical treatment, open biopsy, and significant traumatic injury received within 28 days before the start of study treatment.
* Having active or uncontrolled primary autoimmune hemocytopenia, including autoimmune hemolytic anemia (AIHA), primary immune thrombocytopenia (ITP), etc.
* Patients with evidence or history of bleeding constitution; Or any bleeding event (such as gastrointestinal bleeding) greater than or equal to CTCAE level 3 within 4 weeks before the first dose;
* Subjects who had an arteriovenous thrombosis event within 6 months.
* Subjects who had a history of psychotropic substance abuse and are unable to abstain or have mental disorders;
* Subjects with any severe and/or uncontrolled disease.
* Within one weeks before the first dose, the subjects had received proprietary Chinese medicines with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions;
* Study treatment related: subjects received live or mRNA vaccines within 4 weeks before the first treatment or were scheduled to receive live or mRNA vaccines during the study;
* Participated in clinical trials of other antitumor drugs within 4 weeks before the first dose;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | Baseline up to 104 weeks
  DLT will be defined as toxicities that meet pre-defined severity criteria (according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0), and assessed as having a suspected relationship to study drug.
Adverse events (AE) | Baseline up to 104 weeks
  The occurrence of all adverse events (AE).
Serious adverse events (SAE) | Baseline up to 104 weeks
  The occurrence of all serious adverse events (SAE).
Clinical laboratory abnormalities | Baseline up to 104 weeks
  Incidence of participants with abnormal clinical laboratory test results.

SECONDARY OUTCOMES:
Complete remission rate (CRR)/ Complete remission with incomplete bone marrow recovery rate (CRi) | Baseline up to 104 weeks
  The proportion of patients with tumor hat have a complete response or complete remission with incomplete bone marrow recovery after treatment.
Objective Response Rate (ORR) | Baseline up to 104 weeks
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period.
Undetectable measurable residual disease (U-MRD) ratio of peripheral blood and/or bone marrow | Baseline up to 104 weeks
  Refers to the undetected residual lesions. Flow cytometry was used to detect less than 1 Chronic Lymphocytic Leukemia (CLL) cell (less than 10-4) in 10,000 white blood cells in peripheral blood and/or bone marrow.
Duration of complete remission / complete remission with incomplete bone marrow recovery | Baseline up to 104 weeks
  The time from the date of first achieving CR or CRi to the date of first definite disease progression or death from any cause (whichever occurs first).
Duration of Response (DOR) | Baseline up to 104 weeks
  For all subjects whose best response was partial response (PR), Complete Response (CR), the time from the date of first achieving PR, CR to the date of first definite disease progression or death from any cause (whichever occurs first).
Time to complete remission | Baseline up to 104 weeks
  The time from beginning the treatment to the first achieving complete remission/ complete remission with incomplete bone marrow recovery.
Time to remission (TTR) | Baseline up to 104 weeks
  Time from the beginning of treatment to the first recording of remission (PR or better remission), only the remission population will be analyzed.
Progression Free Survival (PFS) | Baseline up to 104 weeks
  The time from the first dose to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Overall Survival (OS) | Baseline up to 104 weeks
  The time from start of study treatment to date of death due to any cause.
2 years' PFS rate | Baseline up to 104 weeks
  The proportion of patients with progression free survival in 2 years.
2 years' OS rate | Baseline up to 104 weeks
  The proportion of patients achieving overall survival in two years.
Time to reach the maximum plasma concentration (Tmax) | Before the first dose of TQB3702 tablet and target dose of TQB3909 tablet. 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after the first target dose of TQB3909 tablet. The 4th /11th day before dosing with target dose of TQB3909 tablet.
  Time to reach the maximum plasma concentration after dose
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) | Before the first dose of TQB3702 tablet and target dose of TQB3909 tablet. 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after the first target dose of TQB3909 tablet. The 4th /11th day before dosing with target dose of TQB3909 tablet.
  Cmax is the maximum plasma concentration of TQB3909 and TQB3702
Minimum steady-state plasma drug concentration during a dosage interval (Css-min) | Before the first dose of TQB3702 tablet and target dose of TQB3909 tablet. 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24 hours after the first target dose of TQB3909 tablet. The 4th /11th day before dosing with target dose of TQB3909 tablet.
  Cmin is the minimum plasma concentration of TQB3909 and TQB3702.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China